CLINICAL TRIAL: NCT01357395
Title: A Phase 2, Open-Label, Multi-Center Study of Amuvatinib in Combination With Platinum-Etoposide Chemotherapy in Small Cell Lung Cancer Subjects Who Have Not Responded to Standard Treatment or Relapsed After Standard Treatment
Brief Title: A Phase 2, Open-Label Study of Amuvatinib in Combination With Platinum-Etoposide Chemotherapy in Small Cell Lung Cancer
Acronym: ESCAPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-0470-07; 2010-024378-21 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-05-20 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amuvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amuvatinib (Experimental): Amuvatinib 300 mg PO TID + standard-of-care platinum-etoposide
  Interventions: Drug: Amuvatinib

INTERVENTIONS:
Drug: Amuvatinib — Amuvatinib 300 mg PO TID
  Other Names: MP-470

SUMMARY:
The purpose of the study is to evaluate the safety and potential benefit of combination amuvatinib with standard of care chemotherapy treatment (platinum and etoposide) in small cell lung cancer (SCLC) subjects.

DETAILED DESCRIPTION:
Amuvatinib is an oral multi-targeted tyrosine kinase inhibitor which inhibits the mutant forms of c-Kit and PDGFR alpha. It also disrupts DNA repair likely through suppression of Homologous Recombination protein Rad51. In a Phase 1b clinical study in combination with VP-16 and carboplatin, responses in SCLC were observed. In vitro and in vivo data demonstrated amuvatinib synergy with VP-16 thereby further supporting this combination for continued evaluation in clinical trials. Pharmacokinetic data from Phase 1 clinical trials suggest that co-administration of amuvatinib did not alter exposures of standard of care agents VP-16 or carboplatin as measured by overall exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 of age at the time of consent and have histologically or cytologically confirmed SCLC
2. Measurable SCLC per RECIST guideline that meets one of the following:

   * Disease progression by RECIST at anytime during platinum-etoposide (PE) chemotherapy;
   * Relapse by RECIST within 90 days after completing PE chemotherapy;
   * Stable disease by RECIST as best response after at least two (2) ≥ 21-day cycles of PE chemotherapy. The assessment of stable disease should be made at least 2 weeks after the start of the second cycle

   Subjects who received another second-line therapy are eligible if they still fulfill any one of the above three conditions, and all other eligibility criteria
3. Start treatment with the same last regimen (dose and schedule) of first-line PE chemotherapy that they progressed or relapsed on, including any dose reductions because of toxicity, prior to study entry
4. ECOG performance status 0 to 2
5. Adequate organ function
6. Subjects with screening 12-lead ECG with measurable QTc interval of < 450 msec. If QTc ≥ 450 msec, then confirm the reading by evaluating the mean QTc interval of triplicate ECGs.
7. Sign approved informed consent form

Exclusion Criteria:

1. Prior exposure to amuvatinib
2. No longer eligible for first-line PE chemotherapy due to toxicity and the Investigator believes that the risk of retreating with the same PE chemotherapy regimen would outweigh the benefit
3. Ongoing toxicity from prior treatment unless the toxicity has resolved, or in the opinion of the Investigator, is stable and does not compromise the safety of the subject
4. Mixed SCLC and non-small cell lung cancer, or large cell lung cancer
5. Untreated, unstable, or symptomatic brain metastasis
6. Hypersensitivity to amuvatinib, excipients of amuvatinib, or any agent given in association with this trial
7. A life-threatening illness, medical condition or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or interfere with study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05-28 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate (CR or PR) | 3 months

SECONDARY OUTCOMES:
Progression-free survival and overall survival | 6 months
Disease control rate | 6 months
Duration of response | 6 months
Safety and tolerability | 6 months
Amuvatinib and metabolites PK and other biomarkers | 6 months
Amuvatinib PK interactions with platinum-etoposide chemotherapy | 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Poland (5):
  - Wojewódzki Szpital Specjalistyczny, Radom, Masovian Voivodeship
  - Centrum Onkologii - Instytut im. M. Sklodowskiej-Curie w Warszawie, Warsaw, Masovian Voivodeship
  - Wojewódzki Szpital im. Św. Ojca Pio w Przemyślu Oddział Onkologiczny z Pododdziałem Dziennej Chemioterapii, Przemyśl, Podkarpackie Voivodeship
  - Wojewódzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Specjalistyczny Szpital im. Alfreda Sokolowskiego, Szczecin, West Pomeranian Voivodeship